CLINICAL TRIAL: NCT04682808
Title: A Phase I Trial to Evaluate the Tolerability、Pharmacokinetics and Preliminary Antitumor Activity of FCN-338 in Patients With CLL/SLL
Brief Title: A Study of FCN-338 in Patients With Chronic CLL/SLL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fochon Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-338-002
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: BCL-2; CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): FCN-338 will be given orally in ascending doses in patients with relapsed or refractory CLL/SLL , until the maximum tolerated dose or recommended dose is reached. Followed by up to 43 patients enrolled in the expansion cohort at the recommended dose.
  Interventions: Drug: FCN-338

INTERVENTIONS:
Drug: FCN-338 — FCN-338 will be given orally in ascending doses starting at 50 mg QD until the maximum tolerated dose or recommended dose is reached.

SUMMARY:
This study is being done to evaluate the Tolerability、Pharmacokinetics and Preliminary antitumor activity of oral FCN-338 for the treatment of patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), who have failed or are intolerant to one or more lines of established therapy or for whom no other treatment options are available.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase I dose escalation study of Tolerability、Pharmacokinetics and Preliminary antitumor activity of FCN-338 in ascending cohorts to determine the MTD or recommended dose in patients with relapsed or refractory CLL/SLL patients. This is to be followed by a cohort expansion phase at the MTD or recommended oral dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years，no gender limitation；
2. According to the 2018 iwCLL guidelines ，diagnosed as chronic lymphocytic leukemia or small cell lymphoma;
3. Refractory or recurrent CLL/SLL having previously received at least first-line systemic treatment. First-line treatment is defined as the completion of at least 2 cycles of a standard protocol or clinical trial based on current guidelines. Medical record of disease progression after the last treatment failed or remission. According to the 2018 iwCLL guidelines, there are at least one CLL/SLL indications that require treatment. [Refractory definition: treatment failure (without PR) or PD < 6 months after the last chemotherapy); Definition of recurrence: Patients with complete response (CR) or partial response (PR) ≥ 6 months after disease progression (PD)];
4. ECOG Performance Status scored ≤ 1 （Dose Escalation Stage）or ≤ 2（Dose Expansion Stage）；
5. The expected survival is at least 3 months;
6. Adequate hematologic、renal function parameters；
7. If patient have a high risk of developing TLS, The absolute lymphocyte count was ≥ 25× 109/L and there was a lymph node with a maximum diameter ≥ 5 cm assessed by radiology or there was a node with a maximum diameter ≥ 10 cm assessed by radiology ，patient must deal with TLS according to the protocol；
8. For fertile patients: the patient shall consent to effective contraception during the treatment period and for at least 90 days after the last administration of the study treatment, and to receive contraceptive methods such as double-screen contraception, condoms, oral or injectable contraceptives, and intrauterine devices. Male patients should agree to avoid sperm donation;
9. Patients voluntarily signed informed consent;

Exclusion Criteria:

1. The patient's prior antitumor therapy meets one of the following criteria:

   1. Use of other cytotoxic drugs, research drugs or other antitumor drugs within 14 days or 5 half-lives before first receiving study drugs;
   2. Major surgery was performed within 4 weeks prior to the first receiving study drug or had not fully recovered from previous surgery；
   3. Systemic radiotherapy was performed within 28 days prior to the first dose of the study drug, or non-hematological toxicity has not recovered from previous radiotherapy to NCI-CTCAE (version 5.0) level 0-1;
   4. Received anti-tumor monoclonal antibody therapy within 4 weeks before receiving the first study drug;
   5. The toxicity of previous antitumor therapy has not recovered (≥ NCI-CTCAE [version 5.0] level 2), except for hair loss;
   6. Received steroid therapy for antitumor within 7 days before first receiving study drug;
2. Has received allogeneic stem cell transplantation or autologous stem cell transplantation within 6 months prior to first receiving research drug；
3. The biopsy confirmed the transformation to Richter's syndrome；
4. Drug resistance to another bcl-2 family protein inhibitor has occurred (for extend study use only)；
5. Cardiac function and disease meet one of the following conditions:

   1. The prolonged QTc interval has clinical significance, or the screening stage QTc interval is >470ms for women or >450ms for men；
   2. American New York Heart Association (NYHA) grade ≥ 2 congestive Heart failure;
   3. Unstable angina, myocardial infarction, or arrhythmia requiring treatment during screening, Left ventricular ejection fraction (LVEF) <50%; Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmia-causing right ventricular cardiomyopathy, restricted cardiomyopathy, unformed cardiomyopathy);
   4. The investigators determined that the patient's cardiac function can't tolerate to TLS prophylaxis；
6. Patients who have a history of significant renal, neurological, psychiatric, pulmonary, endocrine, metabolic, immunological, cardiovascular or liver diseases that the investigator believes may adversely affect Patients participation in the study；
7. Allergy to the same kind of drugs and excipients used in research；
8. A woman who is pregnant or nursing；
9. Except for adequately treated carcinoma in situ of the cervix, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, and previous malignancies that have been controlled and surgically removed or treated with radical treatment, a history of other active malignancies except for CLL/SLL Within 3 years of the start of the study；
10. Difficulty swallowing, or having malabsorption syndrome or other medical conditions that prevent the absorption of drugs through the intestine；
11. Exhibit other clinically significant uncontrolled conditions, including but not limited to:

    1. Uncontrollable systemic infections (viruses, bacteria, fungi) include viral Hepatitis B (Hepatitis B surface antibody-positive with DNA exceeding 1000 CPS/mL or 1000 IU/ml, or Hepatitis C Virus (HCV) RNA positive)；
    2. An active and uncontrolled autoimmune hemocytopenia lasting 2 weeks or longer, including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura；
12. Systemic diseases that affect patients adherence to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of treatment-related adverse events meeting the criteria for dose limiting toxicities (DLTs) | Cycle 1 (28 days)
To establish the recommended MTD dose and Phase 2 dose (RP2D) of FCN-338 for future clinical trials in patients with advanced CLL/SLL | Up to 24 months
The occurrence of adverse events (AEs) reported in all subjects who received study drug | From enrollment up to 30 days after last dose
The occurrence of treatment-emergent adverse events (TEAs) | From first dose up to 30 days after last dose

SECONDARY OUTCOMES:
Pharmacokinetic variables including maximum plasma concentration (Cmax) | Cycle 1 (28 days)
Pharmacokinetic variables including minimum plasma concentration (Cmin) | Cycle 1 (28 days)
To quantify the last time point with a quantifiable concentration (AUClast) of FCN-338 | Cycle 1 (28 days)
To measure the time to reach the highest plasma concentrations (Tmax) of FCN-338 | Cycle 1 (28 days)
To quantify the terminal half-life (T1/2) of FCN-338 after administration as a single agent | Cycle 1 (28 days)
To quantify the plasma clearance (CL/f) of FCN-338 after administration as a single agent | Cycle 1 (28 days)
To determine the best overall response rate (ORR) by Response Criteria in Solid Tumors (RECIST) v1.1 in subjects with Chronic CLL/SLL | Measured up to 2 years after the last participant has enrolled in the study

CONTACTS AND LOCATIONS:
Overall Officials: Huang Hui Qiang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- SUN YAT-University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No